CLINICAL TRIAL: NCT04387344
Title: Cardiac Modifications in Transthyretin Cardiac Amyloidosis
Brief Title: Morpho-functional Cardiac Modifications in Treated Mutated Transthyretin Cardiac Amyloidosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Messina (Other)
Collaborators: Campisi Mariapaola (Unknown)
Responsible Party: Principal Investigator, Gianluca Di Bella, Associate Professor Cardiovascular Diseases, University of Messina
Other Study IDs: UNIME_CARD_2
Record Dates: First submitted 2020-05-03; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac Amyloidosis (CA) is characterized by a long subclinical phase characterized by deposition of amyloid fibrils in atria, valves and walls of ventricles. Longitudinal dysfunction of the left ventricle (LV) with preserved ejection fraction (EF) is the early phase of CA.

Longitudinal dysfunction mainly involves the LV basal and middle segments with less involvement of the distal segments (apical sparing).

Strain echocardiography (STE) measures myocardial deformation. The technique has been shown to be sensitive for early detection of impaired systolic function and for the study of CA. Additionally, cardiac efficiency (myocardial work) can be derived from myocardial strain data analysis.

In the year 2018, "RNA interferences" (patisiran and inotersen) were included in the list of compassionate therapeutic use programs for exclusive use for the treatment of adult patients with hereditary amyloidosis neuropathy. The aim of our study is to evaluate the morpho-functional modifications with RNA interferences.

DETAILED DESCRIPTION:
Transthoracic echocardiographic images are recorded in the available ultrasound units (Vivid 7 and Vivid 9, GE Ultrasound, Horten, Norways and MyLab - Esaote, Genoa, Italy). The diameters and the wall thicknesses are measured according to the insurance of the American Society of Echocardiography. The images obtained with apical view and in format 4 bedrooms with frame rates (70-80 frames / s) - stored for three cardiac cycles in cine-loop format - will be used for evaluate off-line to evaluate left ventricle deformation in the longitudinal and radial direction, basalelateral, and top segments (post processing) through software already in use and available (Suitestenza, Esaote, Florence, Italy and GE Ultrasound, Horten, Norway).

ELIGIBILITY:
Inclusion Criteria:

* presence of data obtained from historical records of patients who retrospectively met the prescriptive (neurological) criteria and received the prescription of the drugs in question (RNA interferences) having
* Cardiological evaluation (examination ECG, echocardiography) at the time of prescription
* Cardiological evaluation (examination ECG, echocardiography) evaluated six months after therapy,
* Cardiological evaluation (examination ECG, echocardiography) evaluated 12-18 months after therapy,

Exclusion Criteria:

* it wasn't possible to putatively confirm the reasonable shipment of the innovative therapy prescribed
* it wasn't possible to putatively confirm the reasonable shipment of conventional therapy prescribed (background therapy)

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a diagnosis amyloidosis treated with RNA interferences. A diagnosis of cardiac amyloidosis requires left ventricular wall thickness of ≥12 and a positive perugini score (grade 2-3) on technetium-99m(99mTc)-diphosphonate (DPD) or 99mTc-hydroxyl-methylene-diphosphonate (HMDP) bone scintigraphy.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-05-20 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Atrial and Ventricular Walls Dimensions | Change from Baseline Wall Thickness to 18 months
  Measurements (mm) of Interatrial Septum, Ventricular Walls, Coumadin Ridge, Mitro-aortic Lamina, Valves
Change of Atrial and Ventricular Strain | Change from Baseline Atrial and Ventricular Strain to 18 months
  Mean paired change in myocardial strain (percent) by echocardiographic strain-rate imaging (unitless)

SECONDARY OUTCOMES:
Change of Myocardial Work index of Left Ventricle | Change from Baseline Myocardial work to 18 months
  Evaluation of the Global work index (GWI): total work within the area of the LV pressure-strain loops calculated from mitral valve closure to mitral valve opening.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Di Bella, MD, Principal Investigator — University of Messina, Italy
Locations (2):
- Italy (2):
  - Careggi Hospital, Florence
  - Fondazione Policlinico Universitario A. Gemelli IRCCS., Roma

REFERENCES:
- [Result] Di Bella G, Pizzino F, Minutoli F, Zito C, Donato R, Dattilo G, Oreto G, Baldari S, Vita G, Khandheria BK, Carerj S. The mosaic of the cardiac amyloidosis diagnosis: role of imaging in subtypes and stages of the disease. Eur Heart J Cardiovasc Imaging. 2014 Dec;15(12):1307-15. doi: 10.1093/ehjci/jeu158. Epub 2014 Sep 4. PMID 25190073
- [Result] Di Bella G, Minutoli F, Piaggi P, Casale M, Mazzeo A, Zito C, Oreto G, Baldari S, Vita G, Pingitore A, Khandheria BK, Carerj S. Usefulness of Combining Electrocardiographic and Echocardiographic Findings and Brain Natriuretic Peptide in Early Detection of Cardiac Amyloidosis in Subjects With Transthyretin Gene Mutation. Am J Cardiol. 2015 Oct 1;116(7):1122-7. doi: 10.1016/j.amjcard.2015.07.008. Epub 2015 Jul 16. PMID 26253999
- [Result] Di Bella G, Minutoli F, Pingitore A, Zito C, Mazzeo A, Aquaro GD, Di Leo R, Recupero A, Stancanelli C, Baldari S, Vita G, Carerj S. Endocardial and epicardial deformations in cardiac amyloidosis and hypertrophic cardiomyopathy. Circ J. 2011;75(5):1200-8. doi: 10.1253/circj.cj-10-0844. Epub 2011 Mar 17. PMID 21427499
- [Result] Emdin M, Aimo A, Rapezzi C, Fontana M, Perfetto F, Seferovic PM, Barison A, Castiglione V, Vergaro G, Giannoni A, Passino C, Merlini G. Treatment of cardiac transthyretin amyloidosis: an update. Eur Heart J. 2019 Dec 1;40(45):3699-3706. doi: 10.1093/eurheartj/ehz298. PMID 31111153
- [Result] Benson MD, Waddington-Cruz M, Berk JL, Polydefkis M, Dyck PJ, Wang AK, Plante-Bordeneuve V, Barroso FA, Merlini G, Obici L, Scheinberg M, Brannagan TH 3rd, Litchy WJ, Whelan C, Drachman BM, Adams D, Heitner SB, Conceicao I, Schmidt HH, Vita G, Campistol JM, Gamez J, Gorevic PD, Gane E, Shah AM, Solomon SD, Monia BP, Hughes SG, Kwoh TJ, McEvoy BW, Jung SW, Baker BF, Ackermann EJ, Gertz MA, Coelho T. Inotersen Treatment for Patients with Hereditary Transthyretin Amyloidosis. N Engl J Med. 2018 Jul 5;379(1):22-31. doi: 10.1056/NEJMoa1716793. PMID 29972757
- [Result] Adams D, Gonzalez-Duarte A, O'Riordan WD, Yang CC, Ueda M, Kristen AV, Tournev I, Schmidt HH, Coelho T, Berk JL, Lin KP, Vita G, Attarian S, Plante-Bordeneuve V, Mezei MM, Campistol JM, Buades J, Brannagan TH 3rd, Kim BJ, Oh J, Parman Y, Sekijima Y, Hawkins PN, Solomon SD, Polydefkis M, Dyck PJ, Gandhi PJ, Goyal S, Chen J, Strahs AL, Nochur SV, Sweetser MT, Garg PP, Vaishnaw AK, Gollob JA, Suhr OB. Patisiran, an RNAi Therapeutic, for Hereditary Transthyretin Amyloidosis. N Engl J Med. 2018 Jul 5;379(1):11-21. doi: 10.1056/NEJMoa1716153. PMID 29972753